CLINICAL TRIAL: NCT06984783
Title: Visual Health Evaluation of New Designed Blue-blocking Glasses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: TREC2025-KY060
Record Dates: First submitted 2025-04-27; First posted 2025-05-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-01

CONDITIONS: Blue-blocking Glasses
Keywords: Blue-blocking Glasses; Visual fatigue; BUT; CFF; Visual function
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Intervention Model Description: This study used a within-subject design, where each participant completed both experimental conditions in a randomized order.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Group (Experimental): Is a group that will first wear the new type of filtering glasses for one week of observation, followed by one week of observation wearing regular framed glasses. In this trial group, participants will initially perform VDT (Visual Display Terminal) work while wearing the new filtering glasses for at least two hours per day. On the first afternoon, after wearing blue-light-blocking glasses for two hours of near work on VDT, participants will undergo data collection for the trial (including critical flicker fusion frequency (CFF), binocular visual function, computerized refraction, and tests related to dry eye syndrome, etc.), followed by a visual fatigue questionnaire survey after completing the tasks. For a continuous period of one week, participants will wear blue-light-blocking glasses for at least two hours of near work on VDT each day, and on the seventh afternoon, they will undergo another round of data collection and complete the visual fatigue questionnaire survey.
  Interventions: Combination Product: The new type of filtering glasses can efficiently filter out the high-energy blue and green light within a narrow wavelength band.
- B Group (Experimental): Is a trial group that first wears regular framed glasses for one week of observation, followed by one week of observation wearing a new type of filtering glasses. In this trial group, subjects will first engage in VDT (Visual Display Terminal) work wearing regular framed glasses for at least two hours per day. On the afternoon of the first day, after wearing regular framed glasses for two hours of near work with VDT, experimental data will be collected (including CFF, binocular visual function, computerized refraction, and tests related to dry eye syndrome, etc.). After completing the tasks, a visual fatigue questionnaire will be conducted. For a continuous period of one week, subjects will wear blue-light filtering glasses for at least two hours of near work with VDT each day. On the afternoon of the seventh day, experimental data collection and a visual fatigue questionnaire will be conducted again.
  Interventions: Combination Product: The new type of filtering glasses can efficiently filter out the high-energy blue and green light within a narrow wavelength band.

INTERVENTIONS:
Combination Product: The new type of filtering glasses can efficiently filter out the high-energy blue and green light within a narrow wavelength band. — The new type of filtering glasses can efficiently filter out narrow-band high-energy blue and green light.
  Other Names: An efficient narrow-band filtering VDT protective eyewear
  Arms: A Group
Combination Product: The new type of filtering glasses can efficiently filter out the high-energy blue and green light within a narrow wavelength band. — The new type of filtering glasses can efficiently filter out narrow-band high-energy blue and green light.
  Other Names: An efficient narrow-band filtering VDT protective eyewear.
  Arms: B Group

SUMMARY:
With the widespread use of electronic display devices, the potential hazards of blue light have become an important public health issue. The primary assessment and main outcome indicators of this experiment are the evaluation of the protective effects of a new type of filtering glasses on visual fatigue in the human eye. Secondary outcome indicators include tear film break-up time, accommodative facility, and subjective visual fatigue scores. Other outcome measurement indicators include visual function indicators such as accommodation and convergence. Baseline values of the above indicators were measured separately, and then specific numerical values of different indicators were collected after working with VDT devices while wearing the new type of filtering glasses or regular framed glasses. These values were statistically compared and analyzed with the baseline values. The study aims to assess the impact of the new type of filtering glasses on relieving visual fatigue and improving visual function.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult population, regardless of gender 2. Refractive error is less than or equal to -2.5D and both eyes achieve corrected visual acuity of 0.8 or higher. 3. Normal intraocular pressure with no organic pathology. 4. No apparent symptoms of dry eye. 5. Willing to cooperate to complete all the tests. 6. Voluntarily signing the informed consent form.

Exclusion Criteria:

* 1: Individuals with strabismus and amblyopia exist. 2: Suffering from congenital eye conditions such as congenital cataracts or congenital retinal diseases.

  3: Those who have undergone intraocular surgery (such as cataract removal, intraocular lens implantation, etc.).

  4: Individuals with refractive media opacity (such as corneal lesions, lens opacity, etc.).

  5: Abnormal intraocular pressure (IOP) (IOP < 10 mmHg or IOP > 21 mmHg, or a bilateral IOP difference of ≥5 mmHg).

  6: Abnormal intraocular pressure (IOP) (IOP < 10 mmHg or IOP > 21 mmHg, or a bilateral IOP difference of ≥5 mmHg).

  7: Only one eye meets the inclusion criteria. 8: Active corneal infections such as bacterial, fungal, viral, or other acute or chronic anterior segment inflammations.

  9: Currently using medications that may lead to dry eye or affect vision and corneal curvature.

  10: Other ocular conditions, such as dacryocystitis, eyelid disorders and abnormalities, abnormal intraocular pressure, and glaucoma.

  11: Unable to undergo regular eye examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2025-04-18 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Critical flicker fusion frequency | Participants underwent two randomized experimental conditions. For each condition, CFF test was administered at baseline (pre-experiment), post-task on day 1, and post-task on day 7, totaling six completions per participant.
  CFF was measured before and after the task by a flicker fusion frequency detection device to assess changes in the degree of ocular fatigue. To compare the difference in CFF after wearing anti-blue glasses with normal glasses and to evaluate the effect of anti-blue glasses in preventing asthenopia.

SECONDARY OUTCOMES:
Visual fatigue | Participants underwent two randomized experimental conditions. For each condition, visual fatigue questionnaires were administered at baseline (pre-experiment), post-task on day 1, and post-task on day 7, totaling six completions per participant.
  The visual fatigue questionnaire utilized in this study consists of a self-report survey with a total of 19 items. It is designed to comprehensively assess the severity of visual fatigue symptoms, with a scoring system ranging from 1 to 7. Higher scores indicate more severe symptoms, encompassing three primary domains: ocular symptoms, visual discomfort, and psychological aspects triggered by visual fatigue.
Measurement of Accommodative Sensitivity with Flip-Chart Post-VDT Tasks | Participants underwent two randomized experimental conditions. For each condition, flip- chart tests were administered at baseline (pre-experiment), post-task on day 1, and post-task on day 7, totaling six completions per participant.
  This clinical study involves the assessment of accommodative sensitivity for both monocular and binocular vision using a flip-chart immediately following each VDT task. The measurement will quantify the number of optotypes correctly identified within one minute, indicative of the subject's accommodative capacity.
Break up time | Participants underwent two randomized experimental conditions. For each condition, BUT tests were administered at baseline (pre-experiment), post-task on day 1, and post-task on day 7, totaling six completions per participant.
  This clinical study included tear film breakup time measurement using fluorescein sodium stained paper immediately after each VDT task, reflecting tear film stability, and evaluating the degree of dry eye
AC/A Ratio Measurement Post-VDT Tasks | Participants underwent two randomized experimental conditions. For each condition, AC/A ratio test was administered at baseline (pre-experiment), post-task on day 1, and post-task on day 7, totaling six completions per participant.
  This study involves the measurement of the AC/A ratio, which is a critical parameter in binocular vision assessment, reflecting the relationship between accommodation (focus adjustment) and convergence (ocular alignment). The AC/ A ratio will be determined using the prism bar technique, which involve adding lenses to stimulate accommodation and measuring the resulting changes in convergence.
equivalent refraction | Participants underwent two randomized experimental conditions. For each condition, SE test was administered at baseline (pre-experiment), post-task on day 1, and post-task on day 7, totaling six completions per participant.
  This clinical study included testing subjects for equivalent refraction diopters, which can indirectly reflect changes in the degree of myopia in the eye after the use of VDT at close range

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospitol,Capital Medical University, Beijing, Beijing/China, China

IPD SHARING:
Plan to Share IPD: No